CLINICAL TRIAL: NCT05708391
Title: Efficacy and Safety of Concurrent Radiotherapy With Realgar-Indigo Naturalis Formula in the Treatment of Childhood Rhabdomyosarcoma
Brief Title: Radiotherapy Combined With Realgar-Indigo Naturalis Formula (RIF) in the Treatment of Rhabdomyosarcoma(RMS) in Children
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XH-23-001
Record Dates: First submitted 2023-01-18; First posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2022-12

CONDITIONS: Rhabdomyosarcoma, Child
MeSH Terms: conditions — Rhabdomyosarcoma | interventions — Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm: Radiotherapy, Realgar-Indigo naturalis formula (Experimental)
  Interventions: Drug: Realgar-Indigo Naturalis Formulation; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Realgar-Indigo Naturalis Formulation — Radiotherapy: after 4 courses of chemotherapy, radiotherapy was started 13 weeks later. The radiotherapy was performed by three-dimensional conformal intensity modulated radiation (IMRT) technique with a dose of 45-50.4 grey, and radiotherapy was performed 5 times per week for 5-6 weeks.
  Oral administration of Realgar-Indigo naturalis formula from 1 week before radiotherapy to the whole radiotherapy period.
  Dosage: oral, according to body weight, 3 times a day.Because the patient constitution is different, may first start from the half dose, within 3 days gradually increases the dose.In this study, the dosage of Realgar-Indigo naturalis formula (250mg per tablet) was determined according to the patient's weight stage.In each body weight segment, 60 mg/kg realgar-indigo naturalis formula were given according to the upper limit of body weight
Radiation: Radiotherapy — Radiotherapy

SUMMARY:
The goal of this clinical trial]is to evaluate the efficacy, safety and feasibility of radiotherapy combined with Realgar-Indigo naturalis formula（An oral arsenic agent）in the treatment of rhabdomyosarcoma in children. Including the occurrence of adverse events and the improvement of quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group performance status score（ECOG PS）: 0-2, and the expected survival time is ≥3 months;
* At least one measurable lesion according to RECIST version 1.1;
* Postoperative pathological diagnosis of rhabdomyosarcoma, pathological staging of Group II-III patients;
* Patients who have not previously received radiotherapy, have received chemotherapy or whose legal guardian refuses to receive chemotherapy, and may have received surgical treatment for the initial diagnosis;
* Normal major organ function, i.e., meeting the following criteria:

  1. Blood routine examination standards shall meet:(No transfusion within 14 days)

     1. Hemoglobin(HB)≥90g/L;
     2. Absolute Neutrophil Count（ANC）≥1.5×109/L;
     3. Platelet count(PLT)≥80×109/L
  2. Biochemical examination shall meet the following standards:

     1. Bilirubin（BIL）<1.25 times the upper limit of normal (ULN);
     2. Alaninetransaminase(ALT) and aspartate transaminase（AST）<2.5 ULN;
     3. Serum creatinine≤1ULN, endogenous creatinine clearance 50ml/min (Cockcroft-Gault formula)
* The subject voluntarily participates in the study, and the patient or legal guardian signs the informed consent form with the consent of the patient, with good compliance and cooperation in follow-up;
* Patients whose physician believes the treatment will benefit.

Exclusion Criteria:

* Previous or concurrent with other malignancies;
* Persons who have been proved to be allergic to Realgar-Indigo naturalis formula and/or its excipients;
* Has a number of factors affecting oral medication (such as inability to swallow, nausea, vomiting, chronic diarrhea and intestinal obstruction, etc.) ;
* Abnormal coagulation function (international normalized ratio(INR) > 1.5, Activated Partial Thromboplastin Time(APTT) > 1.5 uln) , the patients with bleeding tendency (such as active ulcer lesion in stomach, occult blood in stool (+ +) , black stool and/or hematemesis within 3 months, hemoptysis) or the lesion located near the great vessels;
* Tumors involving the skin and/or pharyngeal mucosa with ulceration;
* Have a history of psychotropic substance abuse and can not quit or have mental disorders;
* patients who had participated in clinical trials of other drugs within 4 weeks;
* The patients whose organ function had not recovered more than 35 days after the previous chemotherapy and could not be treated with the next course of chemotherapy;
* No other anti-cancer treatment may be used during radiotherapy except for the treatment prescribed in the protocol;
* According to the researchers' judgment, there are other patients with concomitant diseases that seriously compromise patient safety or affect the patient's ability to complete the study.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 53 (Estimated)
Dates: Start 2023-01-31 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 1-year
  It refers to the proportion of patients with tumor shrinkage reaching a certain level and maintaining it for a certain period of time, including CR and PR cases.Objective tumor response was assessed using the Response Evaluation Criteria in Solid Tumors (RECIST 1.1 criteria).Subjects must have measurable tumor lesions at baseline, and the efficacy evaluation criteria are divided into complete response (CR), partial response (PR), stable disease (SD) and progressive disease (PD) according to RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Disease Control Rate | 1-year
  Refers to the percentage of CR, PR and SD (≥4 weeks) cases in evaluable patients.
Overall survival | 2-year
  Refers to the time from the date of patient enrollment to death due to any cause.
Quality of life score | 1-year
Adverse events | 1-year
  Observe the adverse events occurring in all subjects during the clinical study